CLINICAL TRIAL: NCT02386280
Title: Prevention of Drug Use in Adolescence: Intervening in Parenting Styles
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Helena Maria Tannhauser Barros, DRA, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AMTEPA
Record Dates: First submitted 2014-12-08; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Substance-Related Disorders
Keywords: Primary Prevention; Substance-Related Disorders; Family
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interviewing for Change of Parenting Styles (Experimental): After measured parental style across the scale, the motivational interviewing will be applied in order to modify the parenting styles of risk for involvement with drug use and maintenance of protective factors. This approach will occur in 5 segments .
  Interventions: Behavioral: Motivational Interviewing for Change of Parenting Styles; Behavioral: Psicoeducation
- Psicoeducation (Sham Comparator): General information about drugs and ways of prevention
  Interventions: Behavioral: Psicoeducation

INTERVENTIONS:
Behavioral: Motivational Interviewing for Change of Parenting Styles
  Arms: Motivational Interviewing for Change of Parenting Styles
Behavioral: Psicoeducation

SUMMARY:
To investigate whether brief motivational intervention is associated with the change of parenting style in parents of teenagers seeking to prevent drug use among their children.

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents aged 10-15 years who call for the service call 132 looking for a program to prevent drug use and accept to participate in the study after reading the Statement of Consent

Exclusion Criteria:

* Be excluded individuals that are experiencing difficulty in answering the questions and those who refuse to participate in the study elucidated by IC

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Measure the reduction risk factors for the use of drugs | 6 months
  The outcome will be measured by the Parenting Styles Inventory

CONTACTS AND LOCATIONS:
Locations (1):
- FUHSPortoAlegre, Porto Alegre, Rio Grande do Sul, Brazil